CLINICAL TRIAL: NCT03365115
Title: Influence of Combined Intrathecal Morphine and Fentanyl in Patients Undergoing Total Knee Arthroplasty
Brief Title: Intrathecal Morphine and Fentanyl for Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201712001
Record Dates: First submitted 2017-11-30; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Knee Arthroplasty
Keywords: spinal anesthesia; morphine; fentanyl; pain; knee
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intrathecal fentanyl (Active Comparator)
  Interventions: Drug: Intrathecal fentanyl
- intrathecal morphine (Active Comparator)
  Interventions: Drug: Intrathecal morphine
- intrathecal morphine and fentantyl (Experimental)
  Interventions: Drug: Intrathecal morphine; Drug: Intrathecal fentanyl

INTERVENTIONS:
Drug: Intrathecal morphine — Intrathecal morphine 100 mcg will be injected.
  Arms: intrathecal morphine; intrathecal morphine and fentantyl
Drug: Intrathecal fentanyl — Intrathecal fentanyl 25 mcg will be injected.
  Arms: intrathecal fentanyl; intrathecal morphine and fentantyl

SUMMARY:
This study is planned to investigate the efficacy of combined infusion of intrathecal morphine and fentanyl in patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled total knee replacement under spinal anesthesia
* ASA I-III

Exclusion Criteria:

* Coagulopathy
* Heart disease
* Liver disease
* Kidney disease
* Infection
* Psychological disorder
* Allergy to bupivacaine
* Allergy to morphine
* Allergy to fentanyl
* Inability to use patient-controlled analgesic device
* Opioids due to chronic pain

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores at 6 hour postoperatively | At 6 hour postoperatively
  Postoperative pain scores will be measured using visual-analogue scale (0:no pain, 10: worst imaginable pain).

SECONDARY OUTCOMES:
Postoperative pain scores at 12 and 24 hour postoperatively | At 12 and 24 hour postoperatively
  Postoperative pain scores will be measured using visual-analogue scale (0:no pain, 10: worst imaginable pain).
Patient-controlled analgesic device requirements | At 6, 12, and 24 hour postoperatively
  The requirements of patient-controlled analgesic device will be measured. Morphine will be used for patient-controlled analgesic device. Total dose of morphine used at 6, 12, and 24 hour postoperatively will be measured.
Number of participants with nausea | At 6, 12, and 24 hour postoperatively
Number of participants with vomiting | At 6, 12, and 24 hour postoperatively
Number of participants with pruritus | At 6, 12, and 24 hour postoperatively
Number of participants with respiratory depression | At 6, 12, and 24 hour postoperatively